CLINICAL TRIAL: NCT07193771
Title: Evaluation of Altitude as an Independent Risk Factor for Mortality in Pediatric Acute Respiratory Distress Syndrome: Influence of Oxygenation, Ventilation, and Hospital Structure in a Multicenter Observational Study.
Brief Title: Altitude and Outcomes in Pediatric ARDS: A Multicenter Study
Acronym: LARed-ALT
Status: Recruiting | Type: Observational
Sponsor: Latin American Pediatric Collaborative Network (Other)
Collaborators: Universidad Nacional de Colombia (Other); Fundación Universitaria de Ciencias de la Salud (Other)
Responsible Party: Sponsor
Other Study IDs: LARED-001
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Distress Syndrome, Pediatric; Altitude Hypoxia; High Altitude Effects
MeSH Terms: conditions — Respiratory Distress Syndrome; Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low Altitude PICUs: Children with PARDS admitted to pediatric intensive care units located at altitudes between 0-1500 meters above sea level.
  Interventions: Other: Geographic Altitude
- Intermediate Altitude PICUs: Children with PARDS admitted to pediatric intensive care units located at altitudes between 1501-2500 meters above sea level.
  Interventions: Other: Geographic Altitude
- High Altitude PICUs: Children with PARDS admitted to pediatric intensive care units located at altitudes between 2501-3500 meters above sea level.
  Interventions: Other: Geographic Altitude
- Very High Altitude PICUs: Children with PARDS admitted to pediatric intensive care units located at altitudes above 3500 meters above sea level.
  Interventions: Other: Geographic Altitude

INTERVENTIONS:
Other: Geographic Altitude — Participants are grouped according to the altitude of the pediatric intensive care unit (PICU) where they are admitted: low altitude (0-1500 m), intermediate altitude (1501-2500 m), high altitude (2501-3500 m), and very high altitude (>3500 m). Altitude is treated as the primary exposure variable. No therapeutic intervention is administered as part of this study.
  Other Names: Altitude Exposure

SUMMARY:
This multicenter observational study will evaluate the association between geographic altitude, availability of critical care resources, and clinical outcomes in children with pediatric acute respiratory distress syndrome (PARDS). Data on demographics, physiology, and hospital structure will be collected from PICUs located at different altitudes worldwide. The study aims to identify gaps in PARDS management and provide recommendations adapted to diverse resource settings.

DETAILED DESCRIPTION:
Pediatric acute respiratory distress syndrome (PARDS) is a major cause of admission and mortality in pediatric intensive care units (PICUs). In high-altitude regions, hypoxemia may be exacerbated, complicating diagnostic interpretation and clinical decision-making. At the same time, variability in the availability of advanced resources-such as mechanical ventilation modes, monitoring systems, and trained personnel-could significantly influence outcomes.

This study will prospectively and retrospectively collect clinical, physiological, and institutional data from pediatric cohorts admitted to PICUs situated at different altitudes worldwide. The analysis will explore how altitude and structural resource differences interact with oxygenation and ventilation parameters to affect patient outcomes. The ultimate goal is to generate evidence that supports context-specific guidelines, reduces inequities in critical care delivery, and strengthens pediatric intensive care practices globally.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month (corrected gestational age) and 18 years.
* Admission to a pediatric intensive care unit (PICU) or facility where mechanically ventilated children are cared for.
* Requirement of invasive mechanical ventilation.
* Diagnosis of pediatric acute respiratory distress syndrome (PARDS) according to PALICC criteria, confirmed within 24 hours before or after endotracheal intubation.

Exclusion Criteria:

* Patients with active perinatal lung disease (e.g., neonatal respiratory distress syndrome, pulmonary hemorrhage, persistent pulmonary hypertension of the newborn, early bronchopulmonary dysplasia, meconium aspiration).
* Patients who have received extracorporeal membrane oxygenation (ECMO) prior to or within the first 24 hours of PARDS diagnosis.
* Patients with pre-established limitation of therapeutic effort (LTE) orders or palliative care directives documented before the initiation of invasive mechanical ventilation.
* Readmissions to the PICU during the study period (only the first episode per patient will be included).

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mechanically ventilated children and adolescents (1 month-18 years) admitted to PICUs at different altitudes worldwide, who fulfill PALICC criteria for PARDS within 24 hours before or after intubation.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | From PICU admission until hospital discharge (up to 90 days)
  Proportion of patients with PARDS who die during hospitalization. Mortality is defined as death during the same hospitalization period in which PARDS was diagnosed.

SECONDARY OUTCOMES:
New morbidity at hospital discharge | From PICU admission until hospital discharge (up to 90 days)
  Presence of new functional morbidity measured using Functional Status Score greater than 2.
Ventilator-free days at 28 days. | 28 days after initiation of invasive mechanical ventilation
  Defined as the number of days a patient is alive and free from invasive mechanical ventilation during the first 28 days after initiation of ventilation. Patients who die within 28 days of initiation will be assigned a value of 0. For survivors, ventilator-free days will be calculated as 28 minus the total number of days on invasive mechanical ventilation during this period.
ICU-free days at 28 days. | 28 days after ICU admission
  Defined as the number of days a patient is alive and not admitted to the ICU during the first 28 days after ICU admission. Patients who die within 28 days of ICU admission will be assigned a value of 0. For survivors, ICU-free days will be calculated as 28 minus the total number of days spent in the ICU during this period.

CONTACTS AND LOCATIONS:
Locations (8):
- Clinica Indisa, Santiago, Chile
- Colombia (5):
  - Hospital Universitario Clinica San Rafael, Bogotá, DC
  - Sociedad de Cirugia de Bogota Hospital de San Jose, Bogotá, DC
  - Fundación HOMI, Bogotá, DC
  - Fundacion Hospital Infantil Los Angeles, Pasto, Departamento de Nariño
  - Clínica UROS S.A, Neiva, Huila Department
- Uruguay (2):
  - Centro Hospitalario Pereira Rossell, Montevideo, Montevideo Department
  - Círculo Católico, Montevideo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tinoco-Solorzano A, Avila-Hilari A, Avellanas-Chavala ML, Montelongo FJ, Velez-Paez J, Nieto Estrada V, Viruez Soto A, Molano Franco D, Castelo Tamayo E, Granda Luna I, Salazar Mendoza A, Mamani Cruz L, Galindo Ayala J, Vasquez-Hoyos P, Maldonado Coronel F, Huanca Payehuanca R, Sanchez Medina JR. Definitions and consensus recommendations on critical care medicine at altitude from the Expert Committee on Critical Care Medicine at altitude of the Pan-American and Iberian Federation of Critical Care Medicine and Intensive Care. Med Intensiva (Engl Ed). 2025 Oct;49(10):502256. doi: 10.1016/j.medine.2025.502256. Epub 2025 Aug 9. PMID 40784821
- [Result] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Result] Molano-Franco D, Masclans Enviz JR, Viruez-Soto A, Gomez M, Rojas H, Beltran E, Nieto V, Aliaga-Raduan F, Iturri P, Arias-Reyes C, Soliz J. Inflammation severity, rather than respiratory failure, is strongly associated with mortality of ARDS patients in high-altitude ICUs. Front Physiol. 2025 Jan 15;15:1520650. doi: 10.3389/fphys.2024.1520650. eCollection 2024. PMID 39882326
- [Result] Jibaja M, Ortiz-Ruiz G, Garcia F, Garay-Fernandez M, de Jesus Montelongo F, Martinez J, Viruez JA, Baez-Pravia O, Salazar S, Villacorta-Cordova F, Morales F, Tinoco-Solorzano A, Ibanez Guzman C, Valle Pinheiro B, Zubia-Olaskoaga F, Duenas C, Garcia AL, Cardinal-Fernandez P. Hospital Mortality and Effect of Adjusting PaO2/FiO2 According to Altitude Above the Sea Level in Acclimatized Patients Undergoing Invasive Mechanical Ventilation. A Multicenter Study. Arch Bronconeumol (Engl Ed). 2020 Apr;56(4):218-224. doi: 10.1016/j.arbres.2019.06.024. Epub 2019 Sep 30. English, Spanish. PMID 31582181
- See also: Related Info — https://www.la-red.net/